CLINICAL TRIAL: NCT00377156
Title: Phase III Randomized Trial of the Role of Whole Brain Radiation Therapy in Addition to Radiosurgery in Patients With One to Three Cerebral Metastases
Brief Title: Stereotactic Radiation Therapy With or Without Whole-Brain Radiation Therapy in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N0574; NCCTG-N0574; ACOSOG-N0574; CDR0000499633 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00653 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer; Cognitive/Functional Effects; Lung Cancer; Metastatic Cancer; Prostate Cancer
Keywords: cognitive/functional effects; tumors metastatic to brain; stage IV breast cancer; stage IV prostate cancer; stage IV non-small cell lung cancer; male breast cancer; recurrent breast cancer; recurrent prostate cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Neoplasm Metastasis; Prostatic Neoplasms; Brain Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms, Male | interventions — Radiotherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients undergo stereotactic radiosurgery (SRS)
  Interventions: Radiation: stereotactic radiosurgery
- Arm II (Experimental): Patients undergo SRS as in arm I. Within 14 days, patients then undergo whole-brain radiotherapy 5 days a week for 2.5 weeks.
  Interventions: Radiation: radiation therapy; Radiation: stereotactic radiosurgery

INTERVENTIONS:
Radiation: radiation therapy — Patients undergo radiation therapy 5 days a week for 2.5 weeks
  Arms: Arm II
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Stereotactic radiation therapy can send x-rays directly to the tumor and cause less damage to normal tissue. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known whether stereotactic radiation therapy is more effective with or without whole-brain radiation therapy in treating patients with brain metastases.

PURPOSE: This randomized phase III trial is studying stereotactic radiation therapy and whole-brain radiation therapy to see how well they work compared with stereotactic radiation therapy alone in treating patients with brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with 1 to 3 cerebral metastases treated with stereotactic radiosurgery with vs without whole-brain radiotherapy.

Secondary

* Compare time to CNS (brain) failure in patients treated with these regimens.
* Compare quality of life, duration of functional independence, and long-term neurocognitive status of patients treated with these regimens.
* Compare post-treatment toxicity in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (18 to 59 vs 60 and over), extracranial disease (controlled for ≤ 3 months vs controlled for > 3 months), and number of brain metastases (1 vs 2 vs 3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo stereotactic radiosurgery (SRS).
* Arm II: Patients undergo SRS as in arm I. Within 14 days, patients then undergo whole-brain radiotherapy 5 days a week for 2.5 weeks.

Quality of life, functional independence, and neurocognitive status are assessed at baseline, at the beginning of each treatment, at weeks 6 and 12, and then at 6, 9, 12, 16, 24 , 36, 48, and 60 months.

PROJECTED ACCRUAL: A total of 238 patients will be accrued for this protocol.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cerebral metastases meeting the following criteria:

  * One to three presumed brain metastases
  * Metastases must be from a histologically confirmed extracerebral site (e.g., lung, breast, prostate)

    * Histologic confirmation may have been from the primary tumor site, from another metastatic site (e.g., osseous metastasis, adrenal metastasis), or from the metastatic brain lesion(s)
  * Each lesion must measure less than 3.0 cm by contrast MRI of the brain performed within the past 21 days
  * Lesions must not be within 5 mm of the optic chiasm or within the brainstem
* Eligibility for treatment with gamma knife or linear accelerator-based radiosurgery confirmed by a radiation oncologist
* No primary germ cell tumor, small cell carcinoma, or lymphoma
* No leptomeningeal metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-2
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

  * Male patients must continue to use contraception for 3 months after the completion of radiotherapy
* No pacemaker or other MRI-incompatible metal in the body
* No known allergy to gadolinium

PRIOR CONCURRENT THERAPY:

* More than 7 days since prior and no concurrent chemotherapy
* No prior cranial radiotherapy
* No prior resection of cerebral metastases
* Concurrent hormonal agents, steroids, and/or anticonvulsants allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Brown, MD, Study Chair — Mayo Clinic
Locations (64):
- United States (60):
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente - Division of Research - Oakland, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Owensboro Mercy Medical Center, Owensboro, Kentucky
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Lowell General Hospital, Lowell, Massachusetts
  - Saint Vincent Hospital at Worcester Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - Immanuel Medical Center, Omaha, Nebraska
  - Seacoast Cancer Center at Wentworth - Douglass Hospital, Dover, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Somerset Medical Center, Somerville, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Cape Fear Valley Medical Center Cancer Center, Fayetteville, North Carolina
  - Coastal Carolina Radiation Oncology Center, Wilmington, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Greenville Cancer Center of the Carolinas (CCOP), Greenville, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
- Canada (4):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Sherbrooke, Quebec

REFERENCES:
- [Derived] Churilla TM, Ballman KV, Brown PD, Twohy EL, Jaeckle K, Farace E, Cerhan JH, Anderson SK, Carrero XW, Garces YI, Barker FG 2nd, Deming R, Dixon JG, Burri SH, Chung C, Menard C, Stieber VW, Pollock BE, Galanis E, Buckner JC, Asher AL. Stereotactic Radiosurgery With or Without Whole-Brain Radiation Therapy for Limited Brain Metastases: A Secondary Analysis of the North Central Cancer Treatment Group N0574 (Alliance) Randomized Controlled Trial. Int J Radiat Oncol Biol Phys. 2017 Dec 1;99(5):1173-1178. doi: 10.1016/j.ijrobp.2017.07.045. Epub 2017 Aug 5. PMID 28939223
- [Derived] Brown PD, Jaeckle K, Ballman KV, Farace E, Cerhan JH, Anderson SK, Carrero XW, Barker FG 2nd, Deming R, Burri SH, Menard C, Chung C, Stieber VW, Pollock BE, Galanis E, Buckner JC, Asher AL. Effect of Radiosurgery Alone vs Radiosurgery With Whole Brain Radiation Therapy on Cognitive Function in Patients With 1 to 3 Brain Metastases: A Randomized Clinical Trial. JAMA. 2016 Jul 26;316(4):401-409. doi: 10.1001/jama.2016.9839. PMID 27458945
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At 34 institutions in North America, patients with 1 to 3 brain metastases were randomized to receive SRS or SRS plus WBRT between February 2002 and December 2013. 70 patients accrued by ACOSOG Z0300 were included in the power calculation and also included for this study.
Groups:
- Arm I (SRS): Patients undergo stereotactic radiosurgery (SRS) received 24 Gy in a single fraction if lesions were less than 2.0cm or 20 Gy if lesions were 2 to 2.9 cm in maximum diameter.
- Arm II (SRS+WBRT): Patients undergo stereotactic radiosurgery (SRS) plus whole-brain radiotherapy (WBRT) received 22 Gy in a single fraction if lesions were less than 2.0cm or 18 Gy if lesions were 2 to 2.9 cm in maximum diameter.>
  > Patients randomly assigned to SRS plus WBRT received 30 GY in 12 fractions of 2.5-Gy WBRT delivered 5 days a week. Whole brain radiotherapy began within 14 days of SRS.
Period: Overall Study
Arm/Group | Arm I (SRS) | Arm II (SRS+WBRT)
Started | 111 | 102
Completed | 63 | 48
Not Completed | 48 | 54
Not completed — Death | 23 | 19
Not completed — Withdrawal by Subject | 16 | 24
Not completed — Had follow-up <90 d | 3 | 6
Not completed — Cancellation | 1 | 0
Not completed — Refused testing | 0 | 1
Not completed — Ineligible | 0 | 1
Not completed — Disability or language problem | 0 | 1
Not completed — Other | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (SRS) | Arm II (SRS+WBRT) | Total
Number analyzed (Participants) | 111 | 102 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (10.4) | 61.4 (10.6) | 60.6 (10.5)
Age, Customized [Count of Participants; unit: Participants]
  18 to 59 | 53 | 44 | 97
  >= 60 | 58 | 58 | 116
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 47 | 104
  Male | 54 | 55 | 109
Region of Enrollment [Number; unit: participants]
  Canada | 23 | 22 | 45
  United States | 88 | 80 | 168

OUTCOME MEASURES:

1. Primary Outcome: Neurocognitive Progression as Measured by the Number of Participants With Cognitive Deterioration by 3 Months
Description: The primary endpoint was cognitive deterioration (progression), defined as a decline of greater than 1 SD from baseline on at least 1 of 7 cognitive tests (all tests are standardized based on published norms and transformed so that higher values represent improved cognition) at the 3-month post-SRS evaluation. The number of participants who experienced cognitive deterioration by 3 months is reported for each arm below. For primary analysis of the 3-month cognitive deterioration endpoint, the Fisher exact 2-group binomial test was used to compare the proportion of evaluable patients with 3-month cognitive deterioration between the 2 groups.
Time Frame: 3 months post radiosurgery
Population: Patients who died prior to the 3-month evaluation, who did not return for the 3-month evaluation or a subsequent evaluation, or who did not complete the required baseline tests were excluded from the analysis population for the primary end point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (SRS) | Arm II (SRS+WBRT)
Number analyzed (Participants) | 63 | 48
Participants | 40 | 44
Statistical Analysis 1: Comparison: Arm I (SRS) vs Arm II (SRS+WBRT); Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Percentage = -28.2, 90% CI 2-sided [-41.9 to -14.4] — Cognitive deterioration, the primary end point in evaluable patients at 3 months, was less frequent after Arm I than Arm II (40/63 [63.5%] vs 44/48 [91.7%],> respectively. The percent difference was -28.2%; 90% CI, -41.9% to -14.4%; P < .001)

2. Secondary Outcome: Number of Participants With Local and Distant Tumor Control up to 3 Months
Description: Number of Participants with Local and Distant Tumor Control up to 3 months is defined as....
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (SRS) | Arm II (SRS+WBRT)
Number analyzed (Participants) | 105 | 95
Participants | 79 | 89
Statistical Analysis 1: Comparison: Arm I (SRS) vs Arm II (SRS+WBRT); Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Percentage = -18.4, 95% CI 2-sided [-29.0 to -7.8]

3. Secondary Outcome: Overall Quality of Life, as Measured by Mean Change From Baseline [3 Month]
Description: Quality of Life was assessed using the Functional Assessment of Cancer Therapy-Brain, for which the range is from 0 to 200 and higher scores indicate better QOL. The Quality of Life (QOL) scores were transformed to a 0- to 100-point scale (with 100 being most favorable), in which a 10-point change was considered clinically significant. Intergroup changes in QOL scores were compared using a 2-sample t test.
Time Frame: From Baseline to 3-Month Evaluation
Population: All patients in the SRS and SRS+WBRT groups that had a baseline and 3-month QOL score were used in this analysis.
Measure: Mean (95% Confidence Interval); unit: QOL score change from baseline points
Groups:
- Arm II (SRS+WBRT): Patients undergo stereotactic radiosurgery (SRS) plus whole-brain radiotherapy (WBRT) received 22 Gy in a single fraction if lesions were less than 2.0cm or 18 Gy if lesions were 2 to 2.9 cm in maximum diameter.>
  >>
  >
  >> Patients randomly assigned to SRS plus WBRT received 30 GY in 12 fractions of 2.5-Gy WBRT delivered 5 days a week. Whole brain radiotherapy began within 14 days of SRS.
Arm/Group | Arm I (SRS) | Arm II (SRS+WBRT)
Number analyzed (Participants) | 65 | 50
QOL score change from baseline points | -0.1 [-4.8 to 4.5] | -12 [-17.5 to -6.6]
Statistical Analysis 1: Comparison: Arm I (SRS) vs Arm II (SRS+WBRT); Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 11.9, 95% CI 2-sided [4.8 to 19.0]

4. Secondary Outcome: Long-Term Neurocognitive Status (Long-Term Cognitive Status), as Measured by Percentage of Long-term Survivors With Cognitive Deterioration at 12 Months
Description: Long-Term Neurocognitive Status > To ascertain in patients with one to three brain metastases whether there is better long-term neurocognitive status in patients who receive SRS alone (Arm A) compared to patients who receive SRS combined with WBRT (Arm B). Long-term survival status is defined as evaluable patients who survived for at least 12 months and had at least one cognitive assessment on or after 365 days.
Time Frame: From baseline to 12 months
Population: Patients who survived for at least 12 months and had at least one cognitive assessment on or after 365 days were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (SRS) | Arm II (SRS+WBRT)
Number analyzed (Participants) | 10 | 18
percentage of participants | 60 | 94.44
Statistical Analysis 1: Comparison: Arm I (SRS) vs Arm II (SRS+WBRT); Test type: Superiority or Other; p = 0.04, Fisher Exact; Mean Difference (Final Values) = -34.4, 95% CI 2-sided [-74.4 to 5.5] — The incidence of cognitive deterioration was less in Arm I than Arm II at 12 months (6/10 [60%] vs 17/18 [94.4%]. The percent difference was -34.4% (95% CI: -74.4% to 5.5%; P = .04)

5. Secondary Outcome: Overall Survival
Description: Overall survival, defined as the time from randomization until death due to any cause, was compared between the groups using stratified log-rank tests.
Time Frame: Up to 5 years
Population: A survival comparison was performed on an intention-to-treat basis using the entire study population.
Measure: Median (Full Range); unit: months
Groups:
- Arm II (SRS+WBRT): Patients undergo stereotactic radiosurgery (SRS) plus whole-brain radiotherapy (WBRT) received 22 Gy in a single fraction if lesions were less than 2.0cm or 18 Gy if lesions were 2 to 2.9 cm in maximum diameter.>>
  >> Patients randomly assigned to SRS plus WBRT received 30 GY in 12 fractions of 2.5-Gy WBRT delivered 5 days a week. Whole brain radiotherapy began within 14 days of SRS.
Arm/Group | Arm I (SRS) | Arm II (SRS+WBRT)
Number analyzed (Participants) | 111 | 102
months | 10.4 [0 to 62.5] | 7.4 [0 to 60.9]
Statistical Analysis 1: Comparison: Arm I (SRS) vs Arm II (SRS+WBRT); Test type: Superiority or Other; p = 0.92, Regression, Cox; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.75 to 1.38]

ADVERSE EVENTS:
Time Frame: Up to 60 months from the start of treatment
Description: All patients that began treatment and were assessed at least once for adverse events are included in this analysis. Adverse Events were collected at weeks 6 and 12 after radiation treatment, and at months 6, 9, 12, 16, 24, 36, 48, and 60 after radiation treatment.
Groups:
- Arm II (SRS+WBRT): Patients randomly assigned to SRS plus WBRT received 30 GY in 12 fractions of 2.5-Gy WBRT delivered 5 days a week. Whole brain radiotherapy began within 14 days of SRS.
Arm/Group | Arm I (SRS) | Arm II (SRS+WBRT)
All-Cause Mortality (participants affected / at risk) | 5/68 | 7/64
Serious Adverse Events (participants affected / at risk) | 8/68 | 11/64
Other Adverse Events (participants affected / at risk) | 45/68 | 53/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (SRS) (N=68) | Arm II (SRS+WBRT) (N=64)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Death (General disorders) | 0 (0) | 3 (6)
Disease progression (General disorders) | 3 (6) | 2 (3)
Fatigue (General disorders) | 1 (2) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Bilirubin increased (Investigations) | 0 (0) | 1 (2)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Central nervous system necrosis (Nervous system disorders) | 1 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Thrombosis (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (SRS) (N=68) | Arm II (SRS+WBRT) (N=64)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (12) | 3 (8)
Arrhythmia supraventricular (Cardiac disorders) | 1 (2) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 1 (2) | 1 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (2)
External ear inflammation (Ear and labyrinth disorders) | 2 (4) | 4 (8)
Hearing loss (Ear and labyrinth disorders) | 1 (2) | 11 (28)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (2)
Eye disorder (Eye disorders) | 0 (0) | 1 (2)
Optic nerve disorder (Eye disorders) | 1 (2) | 0 (0)
Retinopathy (Eye disorders) | 1 (2) | 2 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (6) | 1 (2)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (4)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 1 (2) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (62) | 26 (108)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 11 (28) | 14 (52)
Chest pain (General disorders) | 2 (4) | 0 (0)
Edema limbs (General disorders) | 4 (10) | 0 (0)
Fatigue (General disorders) | 8 (22) | 9 (30)
Gait abnormal (General disorders) | 0 (0) | 1 (2)
Localized edema (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 4 (10)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (2)
Gingival infection (Infections and infestations) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 1 (2) | 1 (2)
Pancreas infection (Infections and infestations) | 1 (4) | 0 (0)
Pneumonia (Infections and infestations) | 3 (6) | 1 (4)
Skin infection (Infections and infestations) | 2 (4) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 5 (12) | 11 (26)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (4)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Amylase increased (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 2 (4)
Bilirubin increased (Investigations) | 1 (2) | 1 (2)
Coagulopathy (Investigations) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (2)
INR increased (Investigations) | 0 (0) | 1 (2)
Leukocyte count decreased (Investigations) | 0 (0) | 2 (8)
Lipase increased (Investigations) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (8) | 2 (8)
Neutrophil count decreased (Investigations) | 1 (2) | 2 (8)
Platelet count decreased (Investigations) | 2 (4) | 3 (8)
Weight gain (Investigations) | 1 (2) | 0 (0)
Weight loss (Investigations) | 2 (4) | 1 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (4) | 5 (12)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 5 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (4) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (10) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (8)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Central nervous system necrosis (Nervous system disorders) | 4 (12) | 3 (10)
Cognitive disturbance (Nervous system disorders) | 14 (36) | 13 (42)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 1 (2) | 3 (6)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 5 (12) | 4 (12)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 16 (51) | 13 (40)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 1 (2)
Seizure (Nervous system disorders) | 4 (10) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 2 (4)
Tremor (Nervous system disorders) | 1 (2) | 0 (0)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (2) | 2 (4)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (17) | 6 (20)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 23 (105) | 40 (162)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hematoma (Vascular disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 3 (6)
Thrombosis (Vascular disorders) | 4 (8) | 1 (2)
Vascular disorder (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes